CLINICAL TRIAL: NCT05923333
Title: Bifidobacterium Infantis Supplementation in Early Life to Improve Immunity in Infants Exposed to HIV: a Randomized, Placebo-controlled, Double-blind Trial
Brief Title: B. Infantis Supplementation to Improve Immunity in Infants Exposed to HIV
Acronym: BifIID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Seattle Children's Hospital (Other); University of Stellenbosch (Other); Institute for Systems Biology (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Washington (Other)
Responsible Party: Principal Investigator, Anna-Ursula Happel, Professor, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 697/2022; R01HD109089 (NIH); PACTR202301748714019 (Registry Identifier: Pan African Clinical Trials Registry)
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Hiv; Vaccine Reaction; Microbial Colonization; Infant Development
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B. infantis Rosell®-33 (Active Comparator): Participants will receive 8 x 109 CFU B. infantis Rosell®-33 per dose (single microbial active ingredient) and carrier material (maltodextrin) for 28 days from day 1-3 of life.
  Interventions: Dietary Supplement: B. infantis Rosell®-33
- Placebo (Placebo Comparator): Participants will receive placebo (containing all materials besides B. infantis Rosell®-33) for 28 days from day 1-3 of life.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: B. infantis Rosell®-33 — B. infantis Rosell®-33 + maltodextrin
  Arms: B. infantis Rosell®-33
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to evaluate the effect of early-life B. infantis Rosell®-33 supplementation in infants exposed to HIV on:

* gut microbiome composition and diversity at 4 weeks of life
* markers of intestinal inflammation and microbial translocation at 4 weeks of life
* Th1 cytokine responses to BCG at 7 weeks and 36 weeks of life

The secondary objectives include to evaluate the effect of B. infantis Rosell®-33 supplementation on:

* longitudinal succession of the gut microbiota composition, diversity and function
* relative and absolute abundance of B. infantis in infant stool during the first 36 weeks of life
* stool metabolome
* T cell subset ontogeny during the first 9 months of life.

Exploratory objectives are to evaluate whether B. infantis Rosell®-33 supplementation improves:

* infant growth
* all-cause morbidity
* neurodevelopment during the first 9 months of life
* antibody responses to early childhood vaccines

DETAILED DESCRIPTION:
Infants who are born to mothers with HIV (exposed but uninfected; iHEU) are at higher risk of morbidity and display multiple immune alterations compared to infants who are HIV-unexposed (iHU). Easily implementable strategies to improve immunity of iHEU, and possibly subsequent health outcomes, are needed. iHEU have altered gut microbiome composition and bifidobacterial depletion, and relative abundance of Bifidobacterium infantis has been associated with immune ontogeny, including humoral and cellular vaccine responses. Therefore, a randomized trial of B. infantis Rosell®-33 versus placebo given during the first month of life in South African iHEU will be conducted.

This is a parallel, randomised, controlled study. Two-hundred breastfed iHEU will be enrolled from the Khayelitsha Site B Midwife Obstetric Unit in Cape Town, South Africa and 1:1 randomised to receive 8 x109 CFU B. infantis Rosell®-33 daily or placebo for the first 4 weeks of life, starting on day 1-3 of life. Infants will be followed over 36 weeks with extensive collection of meta-data and samples.

ELIGIBILITY:
Inclusion Criteria Mother:

* Willing and able to provide signed and dated informed consent form
* 18 years of age or older
* Documented HIV seropositive
* Antiretroviral therapy initiated before the third trimester of pregnancy
* Planning on exclusively breastfeeding the infant for the first 6 months of life

Inclusion Criteria Infant:

* Documented HIV seronegative at birth
* Born at term (completed at least 37 weeks of gestation)
* Birth weight >2.4kgs

Exclusion Criteria:

* Severe illnesses, e.g. Sepsis
* current TB or known household TB contact
* Chronic disorder or medications (other than antiretrovirals and cotrimoxazole prophylaxis) that in the opinion of the investigator would alter immunity
* Pregnancy or delivery complications including birth asphyxia, seizures, sepsis, major congenital anomalies or congenital infections
* Known contraindications to components of the interventional products
* Taking additional probiotics or prebiotics
* Any condition that in the opinion of the investigator would make participation in the trial unsafe

Ages: 0 Days to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome | 4 weeks of age
  Alpha (Shannon) and Beta (Bray Curtis and UniFrac) diversity metrics on the entire microbial communities, assessed by bacterial shotgun metagenomics of infant stool, will be compared between treatment arms
Markers of intestinal inflammation and microbial translocation | 4 - 36 weeks of age
  Concentration of markers of intestinal inflammation and microbial translocation (Lipocalin-2 (Lcn-2), sCD163, I-FABP and LBP measured by ELISA in infant plasma) will be compared cross-sectionally at each time point between groups using Mann-Whitney U tests
BCG vaccine respone | 7 weeks of age
  Frequencies of total net cytokine producing cells in response to stimulation with BCG will be compared between arms.
BCG vaccine respone | 36 weeks of age
  Frequencies of total net cytokine producing cells in response to stimulation with BCG will be compared between arms.

SECONDARY OUTCOMES:
Longitudinal succession in gut microbiota composition, diversity and function | 4 - 36 weeks of age
  Longitudinal multi-omic variation will be visualized using PCoA and tSNE plots, and cross-sectional differences in multi-omic profiles will be assessed using PERMANOVAs.
Stool metabolome | 4 weeks of age
  For cross-sectional metabolite differential abundance analyses, we will use generalized linear regression (continuous dependent variable) and logistic regression (Boolean dependent variable) with an FDR correction.
T cell subsets frequencies | 4 - 36 weeks of age
  T cell subsets frequencies will be compared cross-sectionally between groups

OTHER OUTCOMES:
Presence of total B. infantis and B. infantis Rosell®-33 in stool | 4 - 36 weeks of age
  qPCR will be used to assess whether B. infantis Rosell®-33 colonized.
Infant neurodevelopment milestones | 24 and 36 weeks of age
  Comprehensive neurodevelopment assessment will be conducted, e.g. using the Bayley Scales of Infant and Toddler Development, 3rd edition, or similar assessment tools, and developmental scores compared between the two arms, as well as the proportion of infants passing each developmental area assessed. Higher scores indicate better outcomes.
Infant growth | 4 - 36 weeks of age
  Infant anthropometry will be recorded at each visit to calculate infant length for age (LAZ), weight for age (WAZ) and weight for length (WLZ) Z scores and will be compared between the two arms.
All-cause infectious morbidity | 4 - 36 weeks of age
  Infectious morbidity data will be quantify and compare occurrence of infectious morbidity outcomes between randomisation arms.
Vaccine antibody titres | 4 - 36 weeks of age
  Antibody titres to early childhood vaccines will be assessed and compared by treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Jaspan, MD PHD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Khayelitsha Site B Midwife Obstetric Unit, Cape Town, South Africa

REFERENCES:
- [Derived] Happel AU, Rametse L, Perumaul B, Diener C, Gibbons SM, Nyangahu DD, Donald KA, Gray C, Jaspan HB. Bifidobacterium infantis supplementation versus placebo in early life to improve immunity in infants exposed to HIV: a protocol for a randomized trial. BMC Complement Med Ther. 2023 Oct 18;23(1):367. doi: 10.1186/s12906-023-04208-0. PMID 37853370